CLINICAL TRIAL: NCT01246336
Title: Exploratory Study to Detect Volatile Biomarkers of Idiopathic Parkinson's Disease and Parkinsonism From Exhaled Breath Using a Nanomedical Artificial Olfactory System.
Brief Title: Exploratory Study Using Nanotechnology to Detect Biomarkers of Parkinson's Disease From Exhaled Breath
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Principal Investigator, Ilana Schlesinger, Ilana Schleainger, Rambam Health Care Campus, Rambam Health Care Campus
Other Study IDs: RMB09-0196
Record Dates: First submitted 2010-11-21; First posted 2010-11-23 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Parkinson's Disease; Parkinsonism
Keywords: Parkinson's disease, Parkinsonism; Biomarkers; Exhaled breath; Nanothechnology
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled breath
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with parkinsonism: Patients suffering from Parkinson's disease or parkinsonism
  Interventions: Other: collection of exhaled breath
- Healthy controls: Patients not suffering from Parkinson's disease or any other neurological disorder
  Interventions: Other: collection of exhaled breath

INTERVENTIONS:
Other: collection of exhaled breath — no intervention

SUMMARY:
Parkinson's disease is diagnosed clinically, because biomarkers that may help in diagnosis and differential diagnosis are not yet available. Exhaled breath testing may yield a "breath-print" that can be used to distinguish healthy and diseased states.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinsonism

Exclusion Criteria:

* Severe dementia

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Idiopathic Parkinson's disease and Parkinsonism will be included.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2009-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Nanosensory detection | immediate
  analyze combinations of nanomaterial-based sensors (organically functionalized carbon nanotubes and gold nanoparticles)

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Schlesinger, MD, Principal Investigator — Rambam Health Care Campus